CLINICAL TRIAL: NCT01667367
Title: A Single-center, Single Blind Molecular and Functional Imaging Study to Assess GABAAalpha5 Receptor Expression, Occupancy and Functional Connectivity in the Brains of Individuals With Down Syndrome and Healthy Controls Following a Single Oral Administration of RG1662 or Placebo
Brief Title: A Molecular and Functional Brain Imaging Study in Individuals With Down Syndrome and Healthy Controls Following Single Dose RG1662
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: BP25611; 2012-001301-24 (EudraCT Number)
Record Dates: First submitted 2012-08-14; First posted 2012-08-17 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Volunteer, Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- RG1662 (Experimental)
  Interventions: Drug: RG1662

INTERVENTIONS:
Drug: RG1662 — Single oral dose
  Arms: RG1662
Drug: placebo — Single oral dose
  Arms: Placebo

SUMMARY:
This single-center, single-blind, placebo-controlled, parallel-group study with crossover component will evaluate the GABAAalpha5 receptor expression, occupancy and functional connectivity in the brains of individuals with Down syndrome and healthy controls following single dose RG1662. Participants will receive a single dose of placebo before the imaging session (PET and MRI), and a single dose of RG1662 before the second imaging session.

ELIGIBILITY:
Inclusion Criteria:

Healthy controls and individuals with Down syndrome:

* Male and female adults, 18 to 40 years of age
* Body mass index (BMI) 18 - 40 kg/m2 inclusive
* Females of child-bearing potential and males with female partners of child-bearing potential must agree to use two medically approved methods of contraception, one of which must be a barrier method, for the duration of the study and for 4 months after the last study drug administration
* Clinical laboratory values within normal limits or abnormalities considered not significant by the investigator and sponsor; individuals with thyroid disease may be included in the study provided they are euthyroid and stable on treatment for at least one month prior to screening

Individuals with Down syndrome must also meet the following:

* Diagnosis of Down syndrome confirmed by karyotype; subjects may have free trisomy 21 or Robertsonian translocations; mosaic Down syndrome will be excluded
* Individuals must have a parent or other reliable caregiver who agrees to accompany the inidvidual to all clinic visits, provide information about the individual as required by protocol, and be willing to give informed consent

Exclusion Criteria:

* Regular smoker (>5 cigarettes or equivalent: 3 cigars, 6 cigarillos, 3 pipes per day)
* Concomitant disease or condition or any clinically significant finding at screening that could interfere with, or for which the treatment might interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* Severe head trauma or CNS infections (e.g. meningitis)
* History of epilepsy or seizures other than benign febrile convulsions of childhood
* Any confirmed significant allergic reactions against any drug, anaphylaxis or severe environmental allergies as judged by the investigator
* Positive for hepatitis B, hepatitis C or HIV infection
* Positive urine test at screening or at follow-up for drugs of abuse, or positive alcohol breath test at screening and prior to dosing
* Previous inclusion in research and/or medical protocol involving nuclear medicine, PET or radiological investigations with significant radiation burden (as defined by protocol)
* Pregnant or lactating women
* Individuals with evidence or meeting clinical diagnosis of dementia

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Brain GABAA receptor alpha5 subunit localization/density assessed by positron emission tomography (PET) | approximately 1 day
Brain GABAA receptor alpha5 subunit occupancy following single dose of RG1662 | approximately 1 day
Correlation of RG1662 plasma concentrations and GABAAalpha5 receptor occupancy | approximately 12 months

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 12 months
Resting state functional brain connectivity following a single dose of either RG1662 or placebo, assessed by functional magnetic resonance imaging (fMRI) | approximately 1 day
Functional brain connectivity of individuals with Down syndrome versus healthy controls receiving placebo | approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- London, United Kingdom